CLINICAL TRIAL: NCT05595967
Title: Community Based Health Education for Prevention of Pelvic Floor Dysfunction in Fertile Women in Rural China: Study Protocol for a Non-randomised Cluster Controlled Trial
Brief Title: Community Based Health Education for Prevention of Pelvic Floor Dysfunction in Fertile Women in Rural China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yu Sun, Ph.D., Assistant Director, PKU China Center for Health Economic Research (CCHER), Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PekingUni_Liangshan
Record Dates: First submitted 2022-10-18; First posted 2022-10-27 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Pelvic Floor Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health education intervention (Active Comparator): According the data collected in baseline survey, all participants will be divided into two groups: asymptomatic or mildly symptomatic and severe according the risk level of pelvic floor dysfunction. Intervention for high risk of pelvic floor women focus on emphasizing the need for medical care and access to medical resourced. The first intervention will be performed immediately after baseline survey. The second intervention will be repeated with the first one and performed three months after the first intervention. Both the two session contains modules focusing on heath related knowledge and pelvic floor muscle exercise.
  Interventions: Behavioral: Health education intervention
- Control without intervention (No Intervention): No health education is provided to the participants in the control group so as to investigate the effects of health education. However, materials provided to interventional group will also be sent to the control group after the completion of the study.

INTERVENTIONS:
Behavioral: Health education intervention — Both the two session contains modules focusing on heath related knowledge and pelvic floor muscle exercise. Both two session will be delivered by primary healthcare women workers in small groups (about 20 women per group). The local healthcare workers are responsible for making appointment with each participant through group activities. Each participant will receive a healthy calendar practice to record the number of exercises per day which will be supervised by primary healthcare workers. All healthcare workers are required to attend a full-day workshop organized base on the scheme and teaching materials developed by our research team. The contents of the workshop include: (1) introduction of pelvic floor dysfunction; (2) risk factors and prevention of pelvic floor dysfunction; (3) kegel movement; (4) methods of dealing with severe illness; (5) a standard procedure of group activities or one-on-one activities; (6) skills needed for the delivery of health education intervention.
  Arms: Health education intervention

SUMMARY:
According to the experts in charge of the healthcare department in the Liangshan area, Liangshan is one of the largest Yi inhabited areas in China. Influenced by local culture and production history, most women there are multiparas, with more than one child, and their awareness of postpartum recovery is relatively weak. Therefore, the prevalence and incidence rate of pelvic floor dysfunction diseases is high in the Liangshan area.

In addition, women in the Liangshan area shoulder the responsibility of taking care of family members, farmland, and livestock. They play an important role in family production, which guarantees the opportunity for other family members to go out to work. However, pelvic floor dysfunction can be manifested by persistent pelvic distension, frequent urination, the urgency of urination, difficulty in urination or defecation, and pain or difficulty in sexual intercourse, which decreases the quality of normal life, and the efficiency of production, posing many psychological problems and family contradictions.

There is no research to prove the exact intervention measures that can effectively improve the pelvic floor function of women in Liangshan ethnic minority areas. This study aims to promote the formation of women's healthy living habits and behaviors, improve women's pelvic floor function, and then develop the quality of life and labor output of local women through intervention including health knowledge education and pelvic floor muscle exercise.

ELIGIBILITY:
Inclusion Criteria:

* Married women who are 18-65 years old

Exclusion Criteria:

* Women who are unable to attend the person-to-person health education classes at the first and forth month of the intervention;
* Women who have received pelvic floor muscle training, pelvic floor muscle health education, pelvic floor muscle surgery within one year of the baseline survey;
* Women who are planning pregnancy, pregnant, or have delivered a baby in the past 6 months since the baseline survey;
* Women who are unable to understand the instructions or questions from others.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1139 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-05 (Estimated)

PRIMARY OUTCOMES:
The score of Pelvic Floor Distress Inventory-short form 20 (PFDI-20) | 12 weeks after the start of intervention
  This participant completed questionnaire comprises three subscales with scores ranging from 0 to 100: the Pelvic Organ Prolapse Distress Inventory-6 assessing prolapse symptoms, the ColoRectal-Anal Distress Inventory-8 assessing colorectal/anal symptoms, and the Urinary Distress Inventory-6 assessing urinary symptoms. A higher PFDI-20 score (sum of three subscale scores, range 0-300) indicates a higher symptom burden.
The change in the incidence of pelvic floor dysfunction symptoms | 12 weeks after the start of intervention
  It is defined by the proportion of people who get a PFDI-20 score not equal to 0.

SECONDARY OUTCOMES:
The score of Pelvic Floor Impact Questionnaire-7 (PFIQ-7) | 12 weeks after the intervention
  The Pelvic Floor Impact Questionnaire-7 (PFIQ-7) measuring the changes in condition specific quality of life, which ranges 0-300, with higher scores indicating greater effect.
The score of Prolapse and Incontinence Knowledge Quiz (PIKQ) | 12 weeks after the intervention
  The PIKQ consists of 24 accurate and inaccurate statements related to the epidemiology, pathogenesis, diagnosis and treatment options for urinary incontinence and POP, with which participants were asked if they agreed or disagreed. Each correct response received a score of one, whereas incorrect and "don't know" responses were scored zero. The PIKQ scores (ranging from 0 to 24) were summed and converted to percentages, with higher totals indicating greater pelvic floor knowledge).
Self-reported monthly working days by questionnaire (day) | 12 weeks after the intervention
  This outcome measures the working days of the participants by questionnaire, which indicates whether they are qualified for work.
Self-reported monthly personal income by questionnaire (Yuan) | 12 weeks after the intervention
  This outcome measures the monthly income of the participants by questionnaire, which demonstrates the economic return of their work.

CONTACTS AND LOCATIONS:
Overall Officials: Guoen Liu, PhD, Principal Investigator — Peking University
Locations (1):
- Peking University China Center for Health Economic Research, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data can be provided according to the needs of the researcher, but does not include all personal data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available in 2025
Access Criteria: The data are for research purposes only